CLINICAL TRIAL: NCT05822700
Title: Outcome Of Using Transfixing Hip K Wire ln Developmental Dysplasia Of Hip With Hypoplastic Head And Severe Generalised Ligamentous Laxity
Brief Title: Outcome Of Using Transfixing K Wire ln DDH With Hypoplastic Head And Severe Generalised Ligamentous Laxity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Elbaseet, Professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Developmental Dysplasia of Hip
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Developmental Dysplasia of the Hip
Keywords: Developmental dysplasia of the study; Kirschner wire; Hypoplastic Head; Ligamentous laxity
MeSH Terms: conditions — Developmental Dysplasia of the Hip; Joint Instability | interventions — Bone Wires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- K-wire (Experimental): k wire transfixing hip
  Interventions: Procedure: Kirschner wire

INTERVENTIONS:
Procedure: Kirschner wire — Transfixing femoral head Kirschner wire

SUMMARY:
This study is to evaluate the outcome of using transfixing hip k wire in Developmental dysplastic hip in patients with hypoplastic head and severe generalised ligamentous laxity.

DETAILED DESCRIPTION:
The goal of treatment in developmental dysplasia of the hip (DDH) is to obtain and maintain a stable concentric reduction.

Surgical treatment is done by open reduction through a medial approach or anterolateral approach with pelvic osteotomy,capsulorhaphy, femoral shortening and derotational osteotomy.

Transfixing the femoral head with Kirschner wire during open reduction has long been thought to provide stability to the hip without damaging the femoral head or the acetabulum and to decrease the risk or re-dislocation.

The aim of this study is to assess the effect of transfixing the hip with Kirschner wire during the operative treatment of hip dysplasia in children after the walking age on the final radiological and clinical results and to compare the risks with the benefits of adding this step.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 1 year and younger than 7
2. Patients with hypoplastic head
3. Patients with severe ligamentous laxity (Beighton score ≥ 4)

Exclusion Criteria:

1. Patients younger than 1 year and older than 7 years old.
2. Beighton score < 4
3. Secondary hip dislocation (neuromuscular disorder) as cerebral palsy , myelodysplasia or arthrogryposis.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Modified McKay's criteria | 1 year
  degree of Hip function score

SECONDARY OUTCOMES:
Complications | 1 year
  pain, pin tract infection and recurrent dislocation

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Elbaseet, Professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harsanyi S, Zamborsky R, Krajciova L, Kokavec M, Danisovic L. Developmental Dysplasia of the Hip: A Review of Etiopathogenesis, Risk Factors, and Genetic Aspects. Medicina (Kaunas). 2020 Mar 31;56(4):153. doi: 10.3390/medicina56040153. PMID 32244273
- [Background] Sankar WN, Young CR, Lin AG, Crow SA, Baldwin KD, Moseley CF. Risk factors for failure after open reduction for DDH: a matched cohort analysis. J Pediatr Orthop. 2011 Apr-May;31(3):232-9. doi: 10.1097/BPO.0b013e31820c9b31. PMID 21415680
- [Background] Kamath SU, Bennet GC. Re-dislocation following open reduction for developmental dysplasia of the hip. Int Orthop. 2005 Jun;29(3):191-4. doi: 10.1007/s00264-005-0654-6. Epub 2005 Apr 7. PMID 15815903